CLINICAL TRIAL: NCT00535418
Title: Pre-operative Hormone Therapy for Postmenopausal Women With ER and/or PgR Positive Breast Cancer: An Uncontrolled Phase IIb/III Trial to Assess Optimal Duration of Pre-operative Treatment With Letrozole and to Correlate Clinical Efficacy With Appropriate Surrogate Markers
Brief Title: Optimal Duration of Pre-operative Treatment With Letrozole and to Correlate Clinical Efficacy With Appropriate Surrogate Markers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFEM345EDE01
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Breast cancer; neoadjuvant treatment; treatment duration; Primary hormone receptor positive; breast cancer in postmenopausal women
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

ARMS (1):
- Letrozole (Experimental)
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole
  Other Names: FEM345

SUMMARY:
This study will assess optimal duration of pre-operative treatment with letrozole and to correlate clinical efficacy with appropriate surrogate markers.

ELIGIBILITY:
Inclusion criteria:

1. Female Breast Cancer patients with primary invasive breast cancer, histologically confirmed by core needle biopsy, whose tumors are estrogen (ER) and / or progesterone (PgR) positive (Clinical Stage *T2, T3, T4a,b,c, N0, M0)
2. Patients after menopause
3. Tumor measurable by clinical examination, mammography and ultrasound
4. Adequate bone marrow, renal and hepatic function
5. A life expectancy of at least 6 months.

Exclusion criteria:

1. Prior treatment with aromatase inhibitors or antiestrogens.
2. Uncontrolled endocrine disorders such as diabetes mellitus, confirmed hypo- or hyperthyroidism, Cushing´s Syndrome, Addison´s disease (treated or untreated), Patients with unstable angina, uncontrolled cardiac disease (e.g. Class II or IV New York Heart Association's Functional Classification).
3. Patients with tumors in both breasts, evidence of inflammatory breast cancer or distant metastasis
4. Patients who are eligible for breast conserving surgery.
5. Concomitant anti-cancer treatments such as chemotherapy, immunotherapy/biological response modifiers (BRM's), endocrine therapy (including steroids), bisphosphonate therapy and radiotherapy. Patients who have received HRT will NOT be excluded, provided that HRT is discontinued at least 2 weeks prior to entry into the study.

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2000-06; Primary Completion 2002-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals

REFERENCES:
- [Derived] Krainick-Strobel UE, Lichtenegger W, Wallwiener D, Tulusan AH, Janicke F, Bastert G, Kiesel L, Wackwitz B, Paepke S. Neoadjuvant letrozole in postmenopausal estrogen and/or progesterone receptor positive breast cancer: a phase IIb/III trial to investigate optimal duration of preoperative endocrine therapy. BMC Cancer. 2008 Feb 26;8:62. doi: 10.1186/1471-2407-8-62. PMID 18302747